CLINICAL TRIAL: NCT02281877
Title: Alterations in Skeletal Muscle Gene Expression Following Total Knee Arthroplasty
Brief Title: Alterations in Muscle After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0905
Record Dates: First submitted 2014-10-07; First posted 2014-11-04 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Arthroplasty (TKA); Gene Expression
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Neuromuscular Electrical Stimulation (Experimental): Neuromuscular Electrical Stimulation (NMES) 48 hours after TKA, 5x/week, 2x/day, for 45 minutes/session.
  Standard Rehabilitation Protocol
  Interventions: Procedure: Neuromuscular electrical stimulation (NMES); Behavioral: Standard Rehabilitation Protocol
- Control (Active Comparator): Standard Rehabilitation Protocol
  Interventions: Behavioral: Standard Rehabilitation Protocol

INTERVENTIONS:
Procedure: Neuromuscular electrical stimulation (NMES) — 5x/week, 2x/day, for 45 minutes/session
  Arms: Neuromuscular Electrical Stimulation
Behavioral: Standard Rehabilitation Protocol — Standard physical therapy after TKA

SUMMARY:
The overall goals of this work are: 1) to elucidate alterations in gene expression and downstream protein synthesis 2 weeks after Total Knee Arthroplasty (TKA) to better explain quadriceps muscle atrophy after TKA and 2) understand the mechanisms responsible for improved maintenance of muscle strength with Neuromuscular Electrical Stimulation (NMES) utilization. Furthermore, this investigation seeks to expand previous findings regarding attenuation of strength and functional performance deficits with NMES application to better understand how altered gene expression influences muscle function.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 75 years of age
* Scheduled for unilateral TKA at University of Colorado Hospital
* Diagnosed with osteoarthritis
* Cognitive status that allows patients to consistently comprehend and repeat back directions regarding the details of the study

Exclusion Criteria:

* Neurological, vascular or cardiac problems that significantly limit function
* BMI > 35
* Testosterone supplementation
* Pregnancy
* Anticoagulant therapy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Catabolic gene expression | Change in gene expression from immediately pre surgery to 2 weeks after surgery
  Standard procedures including total RNA isolation, cDNA synthesis, cRNA labeling, microarray hybridization and image acquisition will be performed. Protein content (translation of MAFbx, MuRF1, myostatin) will be analyzed. Total RNA (500 ng) will be reverse transcribed with the iScript cDNA synthesis kit (Bio-Rad, Hercules, CA), and quantitative PCR will be performed using primer sets for genes of interest, reference genes and iQ SYBR Supermix (Bio-Rad) following manufacturer's protocols.

SECONDARY OUTCOMES:
Changes in quadriceps strength | 3 days Pre operative and 2 weeks post operative
  Isometric quadriceps strength will be using a doublet interpolation test performed by research assistants blinded to participants' treatment randomization. Briefly, patients will be seated and stabilized in a HUMAC NORM (Computer Sports Medicine Incorporated, Stoughton, MA) dynamometer with their knee flexed to 60 degrees. After proper warm up, patients will be asked to perform a maximum voluntary isometric contraction of their quadriceps while receiving verbal reinforcement.
Changes in quadriceps size | 3 days Pre operative and 2 weeks post operative
  Peripheral Quantitative Computed Tomography scans of the distal femur will be used to assess the changes in quadriceps muscle morphology quantitatively. The maximal cross-sectional area of the quadriceps will be determined prior to TKA and ~14 days after TKA by manually placing the scanner at a line marked on the vastus lateralis one third of the distance between the greater trochanter and the lateral epicondyle of the femur. The pQCT software will analyze the image and calculate muscle cross-sectional area. A previous investigation by Cramer, et al. validated the pQCT to measurement of muscle cross-sectional area by comparison to MRI and (R2 values of 0.979 and 0.983). In addition, the use of the pQCT to measure muscle cross sectional area had high test-retest reliability, with ICC values of 0.996 and 0.998.
Changes in quadriceps activation | 3 days Pre operative and 2 weeks post operative
  Isometric quadriceps activation testing will be using a doublet interpolation test performed by research assistants blinded to participants' treatment randomization. Briefly, patients will be seated and stabilized in a HUMAC NORM (Computer Sports Medicine Incorporated, Stoughton, MA) dynamometer with their knee flexed to 60 degrees. After proper warm up, patients will be asked to perform a maximum voluntary isometric contraction of their quadriceps while receiving verbal reinforcement. During the contraction, a 2 pulse, 600 µs duration/pulse, supramaximal 100Hz stimulus will be delivered to the muscle to assess whether the subject is indeed maximally contracting the quadriceps muscle and again at rest.
Functional Performance Measures (4 meter walk test, timed up and go, stair climbing test) | 3 days Pre operative and 2 weeks post operative
  The timed Stair Climbing Test (SCT) places a high demand on the quadriceps and therefore measures a higher level of function and, therefore, minimizes the possibility of a ceiling effect. The SCT has been shown to significantly correlate to the Timed Up and Go (TUG). The TUG measures the time it takes a patient to rise from an arm chair (seat height of 46 cm), walk 3 m, turn and return to sitting in the same chair without physical assistance.25 This test has excellent inter-rater (ICC=0.99) and intra-rater reliability (ICC=0.99), as measured in a group of 60 functionally disabled older adults (mean age 80 years).25 The 4 meter Walk Test (4mWT) will be assessed at the fastest safe speed for each participant.
Anabolic Gene Expression | Immediately pre surgery to 2 weeks after surgery
  Standard procedures including total RNA isolation, cDNA synthesis, cRNA labeling, microarray hybridization and image acquisition will be performed. Protein content (translation of mTOR, myogenin, and MyoD) will be analyzed. Total RNA (500 ng) will be reverse transcribed with the iScript cDNA synthesis kit (Bio-Rad, Hercules, CA), and quantitative PCR will be performed using primer sets for genes of interest, reference genes and iQ SYBR Supermix (Bio-Rad) following manufacturer's protocols.
Muscle Fiber Cross-Sectional Area | Immediately pre surgery to 2 weeks after surgery
  Cross sectional area of individual myofibrils taken from the vastus lateralis muscle using immunohistochemical staining and microscopy to determine change in cross sectional area comparing one hour before surgery to two weeks after surgery
Changes in neural cell adhesion molecule (NCAM) concentration | Preop and 2 weeks postop
  NCAM will be assessed by immunohistochemistry with anti-CD56/NCAM antibody (555514; BD Biosciences, San Jose, CA), followed by goat anti-mouse AF555 (A-21127, ThermoFisher). NCAM is a multifunctional cell-surface protein that has been shown to be associated with muscle regeneration, through its roles in neurite outgrowth and synaptic plasticity. NCAM immunohistochemistry will be able to assess 1) denervation status, 2) skeletal muscle response to an intervention, and 3) the capacity for skeletal muscle to improve.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Cheuy, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Univeristy of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado School of Medicine, Aurora, Colorado